CLINICAL TRIAL: NCT00932308
Title: Colorectal Inflammatory Response to a Western-Style Diet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rockefeller University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: PHO-0588
Record Dates: First submitted 2008-12-11; First posted 2009-07-03 (Estimated); Last update posted 2012-02-17 (Estimated); Status verified 2012-02

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Diet, Healthy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Western-style, high-fat, low-calcium diet (WD)
  Interventions: Dietary Supplement: Western-style diet (WD)
- 2 (Active Comparator): Prudent, low-fat, calcium sufficient diet (PD)
  Interventions: Dietary Supplement: Prudent Diet (PD)

INTERVENTIONS:
Dietary Supplement: Western-style diet (WD) — Will comprise of approximately 40% fat, 40% carbohydrates, 20% protein, and 350mg calcium, prepared by the Bionutrition Department using the USDA Nutrient Database.
  Arms: 1
Dietary Supplement: Prudent Diet (PD) — Will contain approximately 20% fat, 60% carbohydrate, 20% protein, and 1100mg calcium; the diets will consist of a 2-day rotating metabolic menu.
  Arms: 2

SUMMARY:
The investigators are involved in a research program to understand how different diets may affect the risk of colorectal polyps and cancer. To that end, the investigators are conducting a study of a western style diet versus a "prudent style" diet in which volunteer subjects are provided a different diet for 2 separate 4 week periods at the Rockefeller University Hospital. During one of these 4 week inpatient periods they receive a Western style diet and during the other 4 week inpatient period they receive a "Prudent style" diet. The investigators will determine changes within the colon as a result of the two different diets. A more detailed description of the study is provided below.

DETAILED DESCRIPTION:
Study subjects participate for about 3 months. During this time, there is one outpatient visit, a 4 week inpatient period, a 4 week outpatient period known as a wash out period and finally another 4 week inpatient period. During the inpatient periods The Rockefeller University Hospital becomes your home the subject must sleep here every night and consume all the food provided. During the screening visit blood and urine samples will be taken and an EKC (electrocardiogram) and a complete physical exam will be done. After enrollment into the study, the first 4 week inpatient period begins. You may continue to go to work or do other activities as long as you eat the diet provided and sleep at the Rockefeller University Hospital. You must eat everything that we give you and you may not substitute or supplement the diet in any way. During each 4 week stay at The Rockefeller University Hospital, there will be three flexible sigmoidoscopies done and biopsies taken of the mucosal lining of the colorectum. This procedure is painless and takes about 5 minutes. In addition, blood and stool samples will be taken every few days for follow-up and research, two 24 hour urine samples will be done on separate days during the hospitalization. Vital signs are measured every day and your weight will be measured three times per week. During the four week wash out period, the subject will return to their home, go about their normal activities and consume their normal diet. The subject will return to The Rockefeller University Hospital for the second 4 week inpatient period. The procedures and laboratory tests are the same during the second inpatient period. The study concludes with the subjects discharge from the RUH.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and post-menopausal healthy female subjects, aged 50-72 years, who have had a colorectal adenoma removed, or have a first or second degree relative with colorectal neoplasia and thus are themselves at risk for colorectal cancer.

Exclusion Criteria:

* Personal history of cancer other than non-melanoma skin cancer within the past 10 years
* History of hereditary non-polyposis colon cancer
* Intestinal malabsorption, inflammatory bowel disease
* Prior gastrointestinal surgery other than appendectomy or surgery of the esophagus
* Any excess bleeding or coagulation disorders
* Subjects taking anti-coagulants, sterol-binding resins, NSAIDs other than aspirin, < 600mg per day, other study medications, or other multiple medications that might, in the view of the study physicians, alter colonic function of inflammation
* Sustained blood pressure > 150/95 mm Hg for three consecutive readings
* Total cholesterol greater than 240mg/dL, triglycerides >600mg, LDL-C > 175
* Subjects with a history of coronary artery disease, with EKG changes consistent with a past myocardial infarction
* HIV positive subjects
* Subjects taking antibiotics, anti-diabetes, hormone replacement therapy, oral, transplanted or injected contraceptives (thyroid hormone therapy is permitted as long as the subjects is euthyroid)
* Subjects consuming a vegetarian diet or a very "prudent diet"

Withdrawal Criteria:

* If a subject is suspected of having taken illicit drugs, the subject will be asked to take a urine test. If positive, the subject will be withdrawn from the study
* The subject takes any medication prescribed without prior approval of the investigator
* Persistent noncompliance with the diets prescribed by the RUH nutritionists

Ages: 50 Years to 72 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2006-09; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
The degree of inflammation in the rectosigmoid epithelium as judged by the density and composition of the cellular infiltration. | Day 1 and Day 28

SECONDARY OUTCOMES:
Expression Profiles of pro- and anti-inflammatory genes in rectosigmoid biopsies as determined by microarray assay and RT-PCR. | Day 1 and Day 28
Selected pro- and anti-inflammatory proteins in rectal biopsies | Day 1 and Day 28
The levels of selected circulating and potential urinary inflammatory markers | Day 27
The concentration of fecal calprotectin | Day -1, 7,14,21 and 27
Changes in bulk fecal and epithelial associated microbiota that may determine changes in colorectal epithelial cell biologic pathways. | Days -1, 7,14,21 and 27

CONTACTS AND LOCATIONS:
Overall Officials: Peter Holt, MD, Principal Investigator — Rockefeller University
Locations (1):
- Rockefeller University, New York, New York, United States